CLINICAL TRIAL: NCT01982227
Title: Monocentric Prospective Pilot Study Evaluating the Value of Indocyanine Green (ICG, Indocyanine Green) During a Surgical Resection of Cancerous Lesions Peritoneal Colorectal Origin.
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1208138; 2012-004314-34 (EudraCT Number)
Record Dates: First submitted 2013-11-06; First posted 2013-11-13 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Colorectal Cancer Metastatic
Keywords: colorectal cancer metastatic; indocyanine green
MeSH Terms: interventions — Indocyanine Green

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients: Patients (Aged 18 to 70 inclusive) with progressive colorectal cancer in intra-abdominal surgery requiring resection +/- Chemotherapy Hyperthermic Intraperitoneal
  Interventions: Drug: indocyanine green

INTERVENTIONS:
Drug: indocyanine green — intravenous injection (0.25mg/kg) of the indocyanine green 24h before the surgery.

SUMMARY:
Between 30% and 40% of patients with colorectal cancer develop metastatic disease intraperitoneally. The optimal treatment of this disease combines surgery and chemotherapy but requires resection of all lesions larger than 2mm.

Indocyanine green has an affinity for tumor tissues and the interest of its use has been demonstrated for the detection of sentinel lymph node and some liver surgeries.

The ability of indocyanine green to detect peritoneal carcinomatosis in humans has never been evaluated.

This study aims to evaluate the diagnostic performance of fluorescence in the detection of malignant cells in peritoneal carcinomatosis of colorectal origin compared with pathological analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patient with progressive colorectal cancer in intra-abdominal surgery requiring resection + / - Chemotherapy Hyperthermic Intraperitoneal
* Aged 18 to 70 inclusive
* Signature information form and consent by the patient

Exclusion Criteria:

* Pregnant women, a urine pregnancy test or blood will be realized within 72 hours before surgery
* Contraindication to surgery
* Diagnosis not confirmed colorectal adenocarcinoma
* Persons major subject of legal protection or unable to consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with progressive colorectal cancer in intra-abdominal surgery requiring resection +/- Chemotherapy Hyperthermic Intraperitoneal
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-03; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Sensitivity (true positive) of the fluorescence ex vivo compared to histological analysis s detected by fluorescence ex vivo | At the end of the surgery
  Sensitivity (true positive) of the fluorescence ex vivo compared to histological analysis s detected by fluorescence ex vivo

SECONDARY OUTCOMES:
Specificity (true negative) of the in-vivo fluorescence compared to histological analysis s detected by fluorescence ex vivo peritoneal cancer index (PCI) score with and without fluorescence | At the end of the surgery
  Specificity (true negative) of the in-vivo fluorescence compared to histological analysis s detected by fluorescence ex vivo PCI score with and without fluorescence
Specificity (true negative) of the in-vivo fluorescence compared to histological analysis s detected by fluorescence ex vivo PCI score with and without fluorescence | At de begining of the surgery
  Specificity (true negative) of the in-vivo fluorescence compared to histological analysis s detected by fluorescence ex vivo PCI score with and without fluorescence

CONTACTS AND LOCATIONS:
Overall Officials: Gabrielle BARABINO, MD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France